CLINICAL TRIAL: NCT05959668
Title: Development of a Patient-reported Outcome to Measure the Health-related Quality of Life of Children, Adolescents and Young Adults With Cystinosis.
Brief Title: Development of Health-related Quality of Life Instrument for Patients With Cystinosis
Acronym: QUALIFY
Status: Recruiting | Type: Observational
Sponsor: Cystinose Stiftung (Other)
Collaborators: Cystinosis Research Network (Unknown); Leben eben! Cystinose-Selbsthilfe e.V. (Unknown)
Responsible Party: Principal Investigator, Julia Hannah Quitmann, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 2205-QUAL-3291
Record Dates: First submitted 2023-05-11; First posted 2023-07-25 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cystinosis
Keywords: Health-related quality of life; Cystinosis; Patient-reported outcome measure
MeSH Terms: conditions — Cystinosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children, adolescents and young adults with cystinosis and their parents: Depending on the patient's age, different HrQoL aspects are more relevant in cystinosis patients and their families. Therefore, a division based on age groups is needed to measure and interpret HrQoL measures successfully:
  Age group stratification will include young patients aged 8-12, 13-17 and 18-26 for a self-reported version and children and adolescents aged 0-4, 5-7, 8-12, 13-17, 18-26 for a parent-reported version.

SUMMARY:
Cystinosis is a rare congenital, inherited metabolic disorder that results in the storage of cystine in the cells of many organs of the body. In the infantile nephropathic form of the disease, only the kidney is initially affected by a loss of function, which progresses if untreated and ends in terminal renal failure by early school age. With the prolonged survival of patients due to medication and renal replacement therapy, further loss of function may occur during the course of the disease, especially in the eyes, muscles, endocrine organs and central nervous system.

The quality of life of children with cystinosis is an under-researched topic. The results of the studies available so far show that the young patients and their families report a reduced quality of life and sometimes behavioral problems.

To date, there are no disease specific patient reported outcome measures (PROMs) to measure the quality of life of patients with cystinosis. The aim of the study is to develop a PROM for this target group in several languages (German, English, Spanish and French) from different countries (Germany, United States, Spain, France). The PROM will focus on quality of life and will be developed for children, adolescents, and young adults including parent-report of parents with children aged 0 to 26 years.

DETAILED DESCRIPTION:
First, a literature review was conducted to identify relevant quality of life topics for the focus interviews. The development of the cystinosis-specific PROM will include three phases with patient recruitment: (1) focus interviews, (2) pilot-test and cognitive debriefing, and (3) field and re-test.

1. Focus interviews with up to 25 parents (of young patients aged 0 to 26) and 15 young patients (ages 8-26) per country (Germany, France, Spain and USA) will discuss aspects relevant to the young patient's quality of life. A pilot instrument version will be developed based on the interviews and then translated into the other project languages according to ISPOR guidelines.
2. The pilot instrument (translated) will be administered to patients and parents along with a cognitive debriefing to assess the comprehensibility, interpretation, and cultural relevance of the items. Up to 200 parents (25-50 per country) and 120 young patients (15-30 per country) will complete the pilot instrument and cognitive debriefing.
3. At least 300 parents (75 per country) and 180 young patients (45 per country) will complete the refined questionnaire as part of a field and re-test.

The questionnaire will be filled out again after two weeks by at least 20% of the patients and parents to assess the test-retest reliability.

The final product will be a psychometrically validated, easy to use, and conceptually appropriate quality of life instrument available in German, English, Spanish, and French for use in research and patient care.

ELIGIBILITY:
In all study phases, patient recruitment follows these inclusion criteria:

Patients will be asked to participate in the study if they meet the following inclusion criteria:

* Children, adolescents, and young adults aged 8-26 years (and at least one of their parents) and further parents only of children aged 0-7
* patients have a confirmed diagnosis of cystinosis
* patients have a sufficient knowledge of the German/ English/ French or Spanish language to participate in focus interviews and complete questionnaires
* the informed consent of legal guardian and assent from the patient (if older than eight years) was given

Exclusion criteria:

* severe cognitive impairment
* other severe illnesses that strongly determine everyday life

Ages: 8 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The participants will be recruited by the Interdisciplinary Cystinosis Clinic in Rosenheim 'RoMed' clinics, the German Cystinosis Foundation, the Cystinosis Research Network, the Asociación Cistinosis Espana, the Necker-Enfants Malades Hospital, the Hospices Civils de Lyon and the VML - Vaincre les Maladies Lysosomales
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interviews with young patients with cystinosis and their parents to identify relevant aspects of disease-specific HrQoL | January 2023 - May 2024
  Semi-structured interviews are conducted to create a pilot test version of the preliminary disease-specific HrQoL tool (QUALIFY). The results of the qualitative analysis will be used to derive an initial item list and response categories of the preliminary questionnaire.
Pilot-test version including a cognitive debriefing to assess the preliminary disease-specific HrQoL tool (QUALIFY) for young people with cystinosis | March 2024 - August 2024
  A pilot-testing of the preliminary version of the QUALIFY questionnaire, including a cognitive debriefing, are performed, so that young patients and parents report on the comprehensibility, completeness, and cultural applicability of the questionnaire from their perspective.
Field-test and of the final version of the disease-specific HrQoL tool (QUALIFY) for young people with cystinosis | September 2024 - April 2025
  A field- and re-test for psychometric assessment of the final version of the QUALIFY questionnaire is performed.

SECONDARY OUTCOMES:
Health related quality of life measured by the chronic-generic DISABKIDS Questionnaire | May 2022 - April 2025
  The 12-item short form of the DISABKIDS Questionnaire is used to assess the HrQoL of children and adolescents with chronic medical conditions from their own as well as their parents' perspectives. The questionnaire consists of three domains: Mental (4 items), social (4 items) and physical (4 items). One composite score can be calculated.
  Higher scores indicate better HrQoL.
Health related quality of life measured by the generic PedsQL™ Generic Core Scales | May 2022 - April 2025
  For the age group 2-4 years, the generic HrQoL of toddlers is assessed via parent report. It consists of 21 items and describes 4 dimensions (Physical Functioning (8 items) Emotional Functioning (5 items) Social Functioning, (5 items), School Functioning (3 items)). The following Scores can be computed: Total Scale Score (21 items); Physical Health Summary Score (8 items); Psychosocial Health Summary Score (15 items).
  The 23-item PedsQL™ Generic Core Scales measure generic HrQoL in children, adolescents, and young adults in self-report as well as proxy report. There are four multidimensional scales (Physical Functioning (8 items) Emotional Functioning (5 items) Social Functioning, (5 items), School Functioning (5 items)) and three summary scores: Total Scale Score (23 items); Physical Health Summary Score (8 items); Psychosocial Health Summary Score (15 items).
  In both versions, scores are transformed to a 0 to 100 scale and higher scores indicate better HrQoL.
Health related quality of life measured by the generic PedsQL™ Infant Scales | May 2022 - April 2025
  The PedsQL™ Infant Scales measure generic HrQoL in infants aged 1-12 and 13-24 months in proxy report.
  The version for infants ages 1-12 months consists of 36 items. There are five multidimensional scales (Physical Functioning (6 items), Physical Symptoms (10 items), Emotional Functioning (12 items) Social Functioning, (4 items), Cognitive Functioning (4 items)).
  The version for infants ages 13-24 months consists of 45 items. There are five multidimensional scales (Physical Functioning (9 items), Physical Symptoms (10 items), Emotional Functioning (12 items) Social Functioning, (5 items), Cognitive Functioning (9 items)).
  In both versions, scores are transformed to a 0 to 100 scale and higher scores indicate better HrQoL. Three summary scores can be calculated: Total Scale Score (all items); Physical Health Summary Score (using items of Physical Functioning and Physical Symptoms); Psychosocial Health Summary Score (Emotional, Social, and Cognitive Functioning items).
Impact of pediatric chronic health condition on parents and the family by the PedsQL™ Family Impact Modules | May 2022 - April 2025
  The 36-item PedsQL™ Family Impact Module describes 8 dimensions: parent self-reported physical functioning (6 items), emotional functioning (5 items), social functioning (4 items), and cognitive functioning (5 items), communication (3 items), worry (5 items), as well as parent-reported family daily activities (3 items) and family relationships (5 items).
  Scores are transformed to a 0 to 100 scale. Higher scores indicate better functioning.
  Three summary scores can be calculated: Total Scale Score (36 items); Parent HrQoL Summary Score (20 items); Family Functioning Score (8 items).
Health related quality of life measured by the newly developed (disease-specific) PROM | September 2024 - April 2025
  The newly developed QUALIFY questionnaire will assess disease-specific HrQoL of young people living wiht cystinosis.
  Higher scores will indicate better HrQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Hannah Quitmann, PD Dr., Study Director — Department of Medical Psychology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany
Locations (1):
- University Medical Center Hamburg-Eppendorf | Center for Psychosocial Medicine | Department of Medical Psychology, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No